CLINICAL TRIAL: NCT01286545
Title: European Ankylosing Spondylitis Infliximab Cohort (EASIC) Follow up Registration Study
Acronym: EASIC registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rheumazentrum Ruhrgebiet (Other)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Braun, Jürgen, Prof. Dr. med, Rheumazentrum Ruhrgebiet, Landgrafenstrasse 15, 44652 Herne
Other Study IDs: EASIC 30505 registry
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; Infliximab; Radiographic progression
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ankylosing spondylitis, long term treatment with infliximab: Patients with ankylosing spondylitis under long term treatment with infliximab within the open label clinical trials EASIC and DIKAS are now followed up in a registration study. No intervention is planned. Patients will be followed up for clinical outcome parameters and for radiographic progression.

SUMMARY:
Long term data on efficacy and safety of anti-TNF treatment with infliximab in patients with ankylosing spondylitis (AS) beyond 5 years is lacking. These data are important because patients with AS usually are younger and withdrawal of anti-TNF therapy in these patients almost always leads to a disease relapse. Furthermore it is still unclear whether long term anti-TNF treatment in AS patients can inhibit radiographic progression. Patients who participated in the EASIC and the DIKAS trial respectively who were treated with infliximab within these studies for 7 and 10 years respectively are followed up by using clinical outcome parameters every 6 months assessing efficacy and safety of long term treatment. Furthermore radiographs of the spine, if done for clinical indication, are analyzed. It is hypothesized that anti-TNF treatment with infliximab is effective and safe over a time period of 9 and 12 years respectively and that long term anti-TNF therapy may inhibit radiographic progression of the spine.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is the most frequent subtype of spondyloarthritides (SpA)(Braun et al.Lancet 2007, 369:1379-90). Treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) is the cornerstone of the treatment of the disease and is widely used to suppress inflammation and ameliorate spinal pain (Zochling et al.:Ann Rheum Dis 2006, 65:442-52). There is evidence that antitumour necrosis factor (TNF) therapy is highly effective in SpA, especially in AS and psoriatic arthritis. Thus, TNF blockers may even be considered as first line treatment in a patient with active AS whose condition is not sufficiently controlled with NSAIDs in the case of axial disease, and sulfasalazine or methotrexate in the case of peripheral arthritis (Zochling et al.:Ann Rheum Dis 2006, 65:442-52). Long-term data on anti-TNF therapy in patients with AS are rather limited. Infliximab in a dosage of 5mg/kg was shown to be efficacious over 5 years, including a short period of withdrawal and readministration (Baraliakos et al.:Arthritis Res Ther 2005, 7: R439-44; Baraliakos et al.:J Rheumatol 2007, 34: 510-5; Braun J et al: Ann Rheum Dis 2008, 67: 340-5). In our EASIC study the investigators have also shown the efficacy and safety of infliximab treatment in patients with AS over 5 years. Long term data for the treatment of AS with etanercept has proven the efficacy as well (Dijkmans B et al.:J Rheumatol 2009, 36: 1256-64). But long term data for efficacy and safety of treatment with anti-TNF therapy beyond a time period of 5 years is lacking. These data on long term treatment are essential for several reasons. At first patients with AS are predominantly of younger age. When taking into account that withdrawal of anti-TNF therapy leads to disease relapse in a very high proportion of patients , anti-TNF therapy in AS patients is most often designed as a continuous therapy on a long term basis. The second reason for the need of long term data beyond 5 years is the ongoing debate whether anti-TNF agents have the potential to inhibit radiographic progression (Baraliakos X et al.:Ann Rheum Dis 2005, 64:1462-6; van der heijde D et al:Arthritis Rheum 2008, 58: 3063-70). Radiographic data on a larger cohort of patients treated with infliximab or other anti-TNF blockers for a long time period could contribute to answer this important question.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of ankylosing spondylitis according to the modified New York criteria
* Participation in the EASIC trial or participation in the DIKAS/TNF bei AS-trial
* Completion of the EASIC extension or the DIKAS trial
* Presence of written informed consent from the patient

Exclusion Criteria:

* None

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ankylosing spondylitis who have completed:
  1. the trials ASSERT, EASIC and EASIC extension (overall 7 years)
  2. the trial DIKAS (overall 10 years)
  and who are still on infliximab or another anti-TNF agent wor who have terminated anti-TNF treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Braun, Prof. Dr., Study Director — Rheumazentrum Ruhrgebiet, Landgrafemstrasse 15, 44652 Herne, Germany
Locations (19):
- Belgium (3):
  - Erasme University Hospital, Brussels
  - Universitair Ziekenhuis, Afdeling Rheumatologie, Ghent
  - University Hospital Leuven, Leuven
- University Central Hospital, Division of Rheumatology, Helsinki, Finland
- France (2):
  - Groupe Hopitalier Cochin, Boulogne
  - Universitat R. Decartes, Hopital Cochin, Paris
- Germany (9):
  - Charité Universitätsmedizin Mitte, Berlin
  - Charité Campus Benjamin Franklin, Berlin
  - Immanuel Krankenhaus Berlin Buch, Berlin
  - Rheumatologie Schlosspark-Klinik, Berlin
  - Rheumapraxis Berlin, Berlin
  - Rheumazentrum Düsseldorf, Universitätsklinik, Düsseldorf
  - Klinik für Immunologie und Rheumatologie der MHH, Hanover
  - Rheumazentrum Ruhrgebiet, Herne
  - Klinikum der Universität München, Rheumaeinheit, München
- Netherlands (2):
  - Academisch Ziekenhuis, Amsterdam
  - University Hospital, Maastricht
- United Kingdom (2):
  - University of Cambridge /Clin Med, Cambridge
  - University of Leeds, Leeds

REFERENCES:
- [Background] Braun J, Sieper J. Ankylosing spondylitis. Lancet. 2007 Apr 21;369(9570):1379-1390. doi: 10.1016/S0140-6736(07)60635-7. PMID 17448825
- [Background] Zochling J, van der Heijde D, Burgos-Vargas R, Collantes E, Davis JC Jr, Dijkmans B, Dougados M, Geher P, Inman RD, Khan MA, Kvien TK, Leirisalo-Repo M, Olivieri I, Pavelka K, Sieper J, Stucki G, Sturrock RD, van der Linden S, Wendling D, Bohm H, van Royen BJ, Braun J; 'ASsessment in AS' international working group; European League Against Rheumatism. ASAS/EULAR recommendations for the management of ankylosing spondylitis. Ann Rheum Dis. 2006 Apr;65(4):442-52. doi: 10.1136/ard.2005.041137. Epub 2005 Aug 26. PMID 16126791
- [Background] Baraliakos X, Listing J, Brandt J, Zink A, Alten R, Burmester G, Gromnica-Ihle E, Kellner H, Schneider M, Sorensen H, Zeidler H, Rudwaleit M, Sieper J, Braun J. Clinical response to discontinuation of anti-TNF therapy in patients with ankylosing spondylitis after 3 years of continuous treatment with infliximab. Arthritis Res Ther. 2005;7(3):R439-44. doi: 10.1186/ar1693. Epub 2005 Feb 21. PMID 15899030
- [Background] Baraliakos X, Listing J, Rudwaleit M, Brandt J, Alten R, Burmester G, Gromnica-Ihle E, Haibel H, Schewe S, Schneider M, Sorensen H, Zeidler H, Visvanathan S, Sieper J, Braun J. Safety and efficacy of readministration of infliximab after longterm continuous therapy and withdrawal in patients with ankylosing spondylitis. J Rheumatol. 2007 Mar;34(3):510-5. Epub 2007 Feb 1. PMID 17299842
- [Background] Braun J, Baraliakos X, Listing J, Fritz C, Alten R, Burmester G, Krause A, Schewe S, Schneider M, Sorensen H, Zeidler H, Sieper J. Persistent clinical efficacy and safety of anti-tumour necrosis factor alpha therapy with infliximab in patients with ankylosing spondylitis over 5 years: evidence for different types of response. Ann Rheum Dis. 2008 Mar;67(3):340-5. doi: 10.1136/ard.2007.075879. Epub 2007 Oct 29. PMID 17967831
- [Background] Dijkmans B, Emery P, Hakala M, Leirisalo-Repo M, Mola EM, Paolozzi L, Salvarani C, Sanmarti R, Sibilia J, Sieper J, Van Den Bosch F, van der Heijde D, van der Linden S, Wajdula J. Etanercept in the longterm treatment of patients with ankylosing spondylitis. J Rheumatol. 2009 Jun;36(6):1256-64. doi: 10.3899/jrheum.081033. Epub 2009 May 1. PMID 19411393
- [Background] Baraliakos X, Listing J, Rudwaleit M, Brandt J, Sieper J, Braun J. Radiographic progression in patients with ankylosing spondylitis after 2 years of treatment with the tumour necrosis factor alpha antibody infliximab. Ann Rheum Dis. 2005 Oct;64(10):1462-6. doi: 10.1136/ard.2004.033472. Epub 2005 Mar 18. PMID 15778240
- [Background] van der Heijde D, Landewe R, Baraliakos X, Houben H, van Tubergen A, Williamson P, Xu W, Baker D, Goldstein N, Braun J; Ankylosing Spondylitis Study for the Evaluation of Recombinant Infliximab Therapy Study Group. Radiographic findings following two years of infliximab therapy in patients with ankylosing spondylitis. Arthritis Rheum. 2008 Oct;58(10):3063-70. doi: 10.1002/art.23901. PMID 18821688
- [Derived] Essers I, van Tubergen A, Heldmann F, Baraliakos X, Braun J, Kiltz U, Boonen A. Do patients with ankylosing spondylitis adapt to their disease? Evidence from a 'then-test' in patients treated with TNF inhibitors. RMD Open. 2015 Nov 17;1(1):e000164. doi: 10.1136/rmdopen-2015-000164. eCollection 2015. PMID 26629367